CLINICAL TRIAL: NCT05999032
Title: The Puerto Rico Asthma Integrated Response Program ("PR-AIR")
Acronym: PR-AIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HL159701 (NIH)
Record Dates: First submitted 2023-05-22; First posted 2023-08-21 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Asthma
Keywords: Pediatric asthma; Community intervention program; Hybrid Type III; Effectiveness and implementation; Home-based intervention; School-based intervention
MeSH Terms: interventions — pleiotrophin

STUDY DESIGN:
Masking Description: There is no masking in this trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-Intensity (Virtual) Intervention Implementation (Active Comparator): During low intensity implementation, families of children with poorly controlled asthma will be referred to the remote version of HARP (HARP-V) and will receive CASE remotely (CASE-V). Children with not well controlled asthma will receive only CASE-V remotely.
  Interventions: Behavioral: CASE in person version (High Intensity Package); Behavioral: CASE-V remote version (Low Intensity Package)
- High Intensity (in-Person) Intervention Implementation (Active Comparator): During high intensity implementation, all interventions are administered in person.
  Specifically, families of children with poorly controlled asthma will receive in-person versions of HARP and CASE. Children with not well controlled asthma will receive an in-person version of CASE only.
  Interventions: Behavioral: CASE and HARP in person (High Intensity package); Behavioral: CASE-V and HARP-V remote version (Low Intensity package)

INTERVENTIONS:
Behavioral: CASE in person version (High Intensity Package) — Controlling Asthma in Schools Effectively (CASE) is a multi-level school-based asthma management program delivered by a Community Health Worker (CHW) that includes 1) staff training involving education on asthma management in school, 2) child-based asthma management education with an emphasis on control of symptoms in the school setting provided in a group setting during the school day, 3) caregiver education after school involving supporting children's asthma control in the school setting, 4), and provision of an Asthma Action Plan (AAP) to the school for child enrollees.
  Arms: Low-Intensity (Virtual) Intervention Implementation
Behavioral: CASE-V remote version (Low Intensity Package) — CASE-V, the low intensity version of CASE, includes similar child and caregiver-based asthma management education that is provided in a remote format with adaptation to integrate technological feature of Zoom. All CASE-V components (for staff, children, and parents) have been adapted to promote engagement (e.g., use of chat and polling function).
  Arms: Low-Intensity (Virtual) Intervention Implementation
Behavioral: CASE and HARP in person (High Intensity package) — Children with "poorly controlled" asthma will receive both the CASE and HARP programs. HARP is a home-visiting program that includes individualized asthma management education and strategies and supplies for environmental remediation. All 3 visits can be conducted by a CHW. The first includes a "walk-through" to identify triggers. Asthma education and self-management strategies are provided using a structured protocol and low-literacy flip-book (English or Spanish). Referrals and advocacy are offered to address asthma management barriers (e.g., communication with landlord/housing re: code violation). The 2nd and 3rd visits include delivery of supplies (e.g., HEPA vacuum, pest gels, mattress covers), instruction for use, review of AAP, and follow-up on environmental control recommendations provided during the 1st visit.
  Arms: High Intensity (in-Person) Intervention Implementation
Behavioral: CASE-V and HARP-V remote version (Low Intensity package) — HARP-V replicates the content delivered in HARP in a remote format. The first session includes a virtual "walk-through" in which the educator uses a structured script and checklist to guide the caregiver through the home and show specific components of the environment (e.g., carpeting, area under the kitchen sink, exhaust fan in bathroom) to identify asthma triggers. Asthma education and self-management strategies are provided using a structured protocol and slide overview based on the HARP flip-book. Supplies for environmental remediation are delivered prior to the 2nd visit. The 2nd and 3rd visit include instruction for use of supplies, review of AAP, and follow-up on recommendations and referrals.
  Arms: High Intensity (in-Person) Intervention Implementation

SUMMARY:
The purpose of this study is to adapt and deliver an evidence-based multi-level intervention to reduce asthma disparities, and that promote and improve population health in the high-burden communities of San Juan, Puerto Rico.

The Puerto Rico-Asthma Integrated Response Program (PR-AIR) will be implemented and evaluated to address pediatric asthma disparities in San Juan, PR, an area of high asthma burden. This study unfolds in two phases: In Phase 1, the researchers will collaborate with community stakeholders to identify needs, barriers and facilitators of PR-AIR implementation. Phase 2 consists of an evaluation of low-intensity (virtual) and high-intensity (in-person) methods of PR-AIR implementation outcomes using the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework and a mixed methods approach.

DETAILED DESCRIPTION:
During the formative evaluation (Phase 1), the researchers will engage community stakeholders (primary caregivers of children with asthma, school personnel, asthma healthcare providers) to help identify, adapt and finalize strategies for PR-AIR implementation. The Consolidated Framework for Implementation Research (CFIR) will be used to identify barriers and facilitators of low-intensity and high-intensity implementation approaches, the Adaptome to guide intervention adaptation to the context of PR, and the CFIR-ERIC matching tool to identify strategies to support but low- and high-intensity implementation packages. Fifteen stakeholders will complete in-depth interviews early in Phase 1, and 16 will participate in two focus groups at the end of Phase 1 prior to the transition to Phase 2, in preparation for trial implementation. A collaborative of community stakeholders will be convened (the PR-AIR CC) to provide input throughout both phases of the trial.

In Phase 2 (Years 2-4) 480 urban children will be enrolled, ages 2-12 (expected retention for full protocol, n = 400) with asthma across 12 areas in San Juan with high asthma burden. Randomization is at the level of targeted geographic area, and data will be collected from groups in each of these areas over time. Individual-level (asthma control, QOL) and community-specific (ED use/hospitalizations, school absence) effectiveness outcomes will be evaluated. All families will participate in both a control (in our case, baseline period for the community indicators) and intervention (active trial). Each target area will begin with a low-intensity (virtual) implementation phase, and transition to a high-intensity implementation phase mid-year. Families enrolled in the first 5 months of the school year will receive the low-intensity intervention package, and those enrolled in the last 5 months of the school year will receive the high-intensity intervention package. Input will be collected throughout each year from community stakeholders about the trial, through in-depth interviews and surveys. Reach, Adoption, Implementation, and Maintenance will be measured using a mixed-methods approach at the end of each trial year (years 2 - 4). Repeated assessments will measure individual-level effectiveness outcomes (asthma control, QOL) at time points linked to the start of intervention participation; at enrollment, end of treatment (EOT; 1 - 2 months after baseline, depending on intervention assignment), and every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Children between the ages of 2 and 12 years old
2. Children must reside in one of the identified catchment areas
3. Children must meet the screening criteria as having not well controlled or poorly controlled asthma

Exclusion Criteria:

1. Children with complex medical conditions

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Child Asthma Control (Individual Level, ages 2-4 years) | Asthma Control will be measured at baseline, End of Treatment (EOT; 1 - 2 months after baseline, depending on intervention assignment), and every 3 months for 1 year.
  Effectiveness of the intervention on child-level asthma control is measured using the Test for Respiratory and Asthma Control in Kids (TRACK). The TRACK is a 5-item measure assessing asthma symptoms and control in young children by caregiver report. Items assessing frequency of various asthma-related events (e.g., breathing problems, quick-relief medication use, etc.) are rated on a Likert-type scale from Not at all (scored 20) to Extremely (scored 0). Scores < 80 suggest child's asthma is not well controlled.
Change in Child Asthma Control (Individual Level, ages 5-11 years) | Asthma Control will be measured at baseline, End of Treatment (EOT; 1 - 2 months after baseline, depending on intervention assignment), and every 3 months for 1 year.
  Effectiveness of the intervention on child-level asthma control is measured using the Childhood Asthma Control Test (cACT). Children answer 4 questions on a 0-3 scale, and caregivers answer 3 questions on a 0-5 scale related to the frequency child's asthma symptoms in the previous 4 weeks. Lower scores indicate worse symptoms. Scores of 19 or less suggest asthma is not well controlled.
Change in Child Asthma Control (Individual Level; ages 12 and up) | Asthma Control will be measured at baseline, End of Treatment (EOT; 1 - 2 months after baseline, depending on intervention assignment), and every 3 months for 1 year.
  Effectiveness of the intervention on child-level asthma control is measured using the Asthma Control Test. Youth ages 12 and up complete 5-items related to their asthma on Likert-type scales ranging from 1-5, with lower scores indicating more severe symptoms. A cutoff score <19 indicates suboptimal asthma control; scores <=15 suggest poorly controlled asthma.
Health Care Utilization-ED visits (Community Level) | 12 months pre- and post-intervention year
  Health care utilization will be assessed by community-level rates of Emergency Department visits of children within the targeted geographic area. Obtaining utilization rates in this way will help the researchers to assess effectiveness of the intervention on the community level.
Health Care Utilization-Hospitalizations (Community Level) | 12 months pre- and post-intervention year
  Effectiveness of the intervention on the community level. Health care utilization will be assessed by community-level rates of hospitalizations in children within the targeted geographic area.
Health Care Utilization-Urgent Care Visits (Community Level) | 12 months pre- and post-intervention year
  Effectiveness of the intervention on the community level. Health care utilization will be assessed by community-level rates of urgent care visits in children within the targeted geographic area.

SECONDARY OUTCOMES:
Asthma-related Quality of Life (QoL) (Individual Level) | Asthma-related QOL will be measured at baseline, End of Treatment (EOT; 1 - 2 months after baseline, depending on intervention assignment), and every three months for 1 year.
  Effectiveness on child-level quality of life (QOL) will be measured by the Pediatric Asthma Quality of Life Questionnaire (PAQLQ). The instrument consists of 23 items related to limitation across three domains (activity limitation, symptoms and emotional function). Each item is rated 1-7 on a Likert scale, with lower numerical responses indicating greater impairment.
School Absences (Community Level) | 12 months pre- and post-intervention year
  Community-level school absences will be assessed by attendance data (i.e., number of school absences) from the schools in the targeted area that correspond to each "step" in the wedge of the study design.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Koinis Mitchell, PhD, Principal Investigator — Rhode Island Hospital; Elizabeth L McQuaid, PhD, ABPP, Principal Investigator — Rhode Island Hospital; Ligia Chavez, PhD, Principal Investigator — University of Puerto Rico
Locations (2):
- Rhode Island Hospital, Providence, Rhode Island, United States
- Medial Sciences Campus, University of Puerto Rico, San Juan, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Following the NIH data sharing policy (2015), within one year of completion of the studies and dissemination of primary study results, public-use analysis datasets will be made available to the public, along with the final version of the study protocol, data dictionaries, and brief instructions. De-identification for the analysis datasets will follow published guidelines for "limited access data sets" funded by NHLBI (Geller et al., 2004).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available within roughly one year of completion of the studies and dissemination of primary study results and will be available for 10 years following the completion of the study.
Access Criteria: Once they become available, researchers requesting the data would follow the PR-AIR data request procedures. We will make the data available to potential users only under a NIH-approved data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant in any way; (2) a commitment to securing the data using appropriate information security that is compliant with the most recent federal guidelines that are outlined by our information security protocol; and (3)a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733
- [Background] CFIR Research Team. Strategy Design [Web]. Consolidated Framework for Implementation Research; 2019 [Available from: https://cfirguide.org/choosing-strategies/ accessed 22 November 2019.
- [Background] Chambers DA, Norton WE. The Adaptome: Advancing the Science of Intervention Adaptation. Am J Prev Med. 2016 Oct;51(4 Suppl 2):S124-31. doi: 10.1016/j.amepre.2016.05.011. Epub 2016 Jun 28. PMID 27371105
- [Background] Waltz TJ, Powell BJ, Fernandez ME, Abadie B, Damschroder LJ. Choosing implementation strategies to address contextual barriers: diversity in recommendations and future directions. Implement Sci. 2019 Apr 29;14(1):42. doi: 10.1186/s13012-019-0892-4. PMID 31036028
- [Background] Murphy KR, Zeiger RS, Kosinski M, Chipps B, Mellon M, Schatz M, Lampl K, Hanlon JT, Ramachandran S. Test for respiratory and asthma control in kids (TRACK): a caregiver-completed questionnaire for preschool-aged children. J Allergy Clin Immunol. 2009 Apr;123(4):833-9.e9. doi: 10.1016/j.jaci.2009.01.058. PMID 19348922
- [Background] Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R. Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy Clin Immunol. 2007 Apr;119(4):817-25. doi: 10.1016/j.jaci.2006.12.662. Epub 2007 Mar 13. PMID 17353040
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Juniper EF, Guyatt GH, Feeny DH, Ferrie PJ, Griffith LE, Townsend M. Measuring quality of life in the parents of children with asthma. Qual Life Res. 1996 Feb;5(1):27-34. doi: 10.1007/BF00435966. PMID 8901364